CLINICAL TRIAL: NCT03000842
Title: Effects of Transcutaneous Vagal Nerve Stimulation (tVNS) on Blood Pressure, Heart Rate and Autonomic Control in Hypertensive Subjects
Brief Title: Effects of Transcutaneous Vagal Nerve Stimulation on Hemodynamics Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 5260/16
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: autonomic control; transcutaneous vagal nerve stimulation; transauricular vagal nerve stimulation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Subjects (Experimental): transcutaneous vagal nerve stimulation
  Interventions: Device: transcutaneous vagal nerve stimulation on; Device: transcutaneous vagal nerve stimulation off
- Hypertensive Subjects (Experimental): transcutaneous vagal nerve stimulation
  Interventions: Device: transcutaneous vagal nerve stimulation on; Device: transcutaneous vagal nerve stimulation off

INTERVENTIONS:
Device: transcutaneous vagal nerve stimulation on — electrical current on positioned in the ear to estimate vagal branch of auricular nerve
Device: transcutaneous vagal nerve stimulation off — an electrical current off positioned in the ear to estimate vagal branch of auricular nerve

SUMMARY:
The vagal stimulation is a promising therapy for a lot of disorders as well as hemodynamic regulatory way. In order to minimize the harm of a surgery chip implantation, actually it was developing a non-invasive device that is able to stimulate the auricular branch of vagal nerve. It has been shown that trans-auricular vagal stimulation (tVNS) causes direct stimulation of the vagal nerve. However, there are still no strong evidences about it actions regarding the autonomic modulation. The aim of this study is to evaluate effects of tVNS on heart rate, blood pressure and the autonomic control in healthy and hypertensive subjects, at rest and after orthostatic position

ELIGIBILITY:
Normotensive group Inclusion Criteria:

* healthy volunteers
* sign the consent term

Normotensive group Exclusion Criteria:

* smokers
* alcoholism
* drug treatment
* skin lesion in the ear region
* chronic or acute diseases
* pregnancy
* be participating in another research protocol
* high performance athletes
* recent surgery
* vaso-vagal syndrome

Hypertensive group Inclusion Criteria:

* hypertensive diagnosis (with or without anti-hypertensive drugs treatment) or
* ambulatory blood pressure monitoring (ABPM) >130/85
* sign the consent term

Hypertensive group Exclusion Criteria:

* smokers
* alcoholism
* beta-blockers treatment
* skin lesion in the ear region
* associated diseases
* pregnancy
* be participating in another research protocol
* high performance athletes
* recent surgery
* vaso-vagal syndrome

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Autonomic control response to transcutaneous vagal nerve stimulation | 40 minutes
  sympathetic and parasympathetic response to non-invasive vagal nerve stimulation

SECONDARY OUTCOMES:
Blood pressure changes to transcutaneous vagal nerve stimulation | 40 minutes
  systemic response to non-invasive vagal nerve stimulation
Heart Rate changes to transcutaneous vagal nerve stimulation | 40 minutes
  cardiac response to non-invasive vagal nerve stimulation